CLINICAL TRIAL: NCT00197197
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group Study to Compare the Efficacy and Safety of GW873140 400mg BID in Combination With a Ritonavir-containing Optimized Background Therapy (OBT) Regimen Versus Placebo Plus OBT Over 48 Weeks.
Brief Title: Study Of Chemokine Coreceptor 5 (CCR5) Antagonist GW873140 In R5/X4-Tropic Treatment-Experienced HIV-Infected Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to hepatoxicity of compound
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCR104458
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infection
Keywords: HIV-1 GW873140 CCR5 antagonist treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — aplaviroc

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: GW873140

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the CCR5 antagonist GW873140 or placebo in combination with an optimized background regimen in treatment-experienced HIV-infected subjects with R5/X4-tropic virus

ELIGIBILITY:
Inclusion criteria:

* HIV-infected.
* Screening viral load at least 5000copies/mL.
* R5/X4-tropic virus at screening.
* Total prior antiretroviral experience of at least 3 months.
* Documented resistance to at least one drug in each of the following classes: nucleoside reverse transcriptase inhibitors (NRTI), non-nucleoside reverse transcriptase inhibitors (NNRTI), and protease inhibitors (PI), stable antiretroviral regimen (or no antiretroviral treatment) for at least 4 weeks before screening.
* Able to receive a ritonavir-boosted protease inhibitor during treatment studies.
* Women of childbearing potential must use specific forms of contraception.

Exclusion criteria:

* Acute laboratory abnormalities.
* History of pancreatitis or hepatitis, hepatitis B or hepatitis C coinfection, or any chronic liver disease. Screening liver function tests will be used to determine eligibility.
* R5-tropic only.
* X4-tropic only.
* non-phenotypeable virus at screening.
* Changes to antiretroviral therapy from 4 weeks prior to screening until Day 1 of treatment study.
* Pregnancy or breastfeeding women.
* Recent participation in an experimental drug trial.
* Prior use of a CCR5 or CXCR4 antagonist.
* Significant ECG abnormalities or significant history of active pancreatitis, hepatitis, opportunistic infections, malabsorption disorders, cancer, or severe illness.
* Current use of certain medications may exclude participation in this study.
* Additional qualifying criteria and laboratory test requirements to be assessed by study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
HIV viral load response at 24 and 48 weeks. | 24 and 48 weeks

SECONDARY OUTCOMES:
Safety and tolerability, change in T-cell count, disease progression, viral resistance,tropism at failure, pharmacokinetics, health outcomes.Liver tests will be done every 2 weeks for 24 weeks. | every 2 weeks for 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Ph.D., Study Director — GlaxoSmithKline
Locations (12):
- United States (11):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Brussels, Belgium